CLINICAL TRIAL: NCT00425217
Title: The Use of Rituximab in the Treatment of Idiopathic Membranous Nephropathy
Brief Title: Rituximab in Membranous Nephropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 627-04
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
Membranous glomerulopathy (MN) is a common immune-mediated glomerular disease and the leading cause of nephrotic syndrome in Caucasian adults. 1 Because of its frequency, it remains the second or third cause of end-stage renal disease caused by a primary glomerulonephritis. 2 At presentation, 70% to 80% of patients have the nephrotic syndrome. 1, 3, 4 Proteinuria greater than 2.0 grams per day is found in > 80% of patients at presentation, with greater than 10 grams found in as many as 30%. 5 The disease affects patients of all ages, but it is most often diagnosed in middle age with the peak incidence during the fourth and fifth decades of life. There is close to a two-to-one predominance of males to females diagnosed with the disease. Idiopathic MN affects all races. Current therapeutic options include corticosteroids alone or in combination with alkylating agents, cyclosporin A, and mycophenolate mofetil. The most widely recognized, and best-validated regimen is combination therapy with corticosteroids and an alkylating agent, but its use is associated with significant adverse effects. Recent meta-analysis confirmed that present day treatments are far from ideal 6 Thus, it should not come as a surprise that the outcome of MN has not substantially improved over the past 30 years, and up to 40% of patients still progress to end-stage renal failure. 7 Like in other glomerular diseases the amount of protein in the urine correlates well with long term prognosis. Thus, this parameter has been used in previous studies, and will be used in this study, as the primary indicator of effectiveness of therapy. We proposed to do a pilot study to test the hypothesis that selective B lymphocyte depletion will result in disappearance of pathogenic antibodies and induction of remission of the nephrotic syndrome in patients with idiopathic membranous nephropathy. Our population will be 10 adults. The study will be conducted between our Nephrology Divisions at Mayo Clinic Rochester, Jacksonville, and Scottsdale. We will enroll patients with a GFR 25 ml/min as estimated by creatinine clearance and proteinuria > 4g/24h, while receiving an ACEI or ARB and with BP controlled of < 130/80 mmHg. Patients will receive Rituximab 1g on Day 1 and 15. Patients followed for 1 years following completion of treatment. The primary outcome will be change in urinary protein excretion at 6 months. Secondary outcomes will be changes in serum albumin, serum lipid?s profile, the number of partial remissions, time to remission, and incidence of relapses. We will also perform a pharmacokinetic study to evaluate the effect of proteinuria on the bio-availability and effects of the drug.

DETAILED DESCRIPTION:
There is convincing evidence from both experimental and human studies that MN is mediated by the deposition of IgG antibodies in the subepithelial aspect of the GBM. More debatable, is the mechanism(s) of deposition of these antibodies in that location. Given the key role of IgG antibodies in MN, it is reasonable to postulate that suppression of antibody production by depleting B cells and/or plasma cells may improve or even resolve the glomerular pathology as reflected by a reduction in proteinuria. There is evidence that this strategy is effective in the treatment of other antibody-mediated diseases and preliminary studies in MN are promising. Data from animal studies suggest that immune deposition resulting from B cell activation promote injury to the glomerular filtering barrier and proteinuria.103 In humans, as discussed above, there is evidence that therapy directed against B cells, e.g. cyclophosphamide, is effective in MN. Cyclophosphamide has striking direct effects on B cell function, and suppresses the secretion of immunoglobulins.104 Thus, a case could be made for using an agent capable of depleting B cells, and therefore halting the production of nephrotoxic immunoglobulins. This approach could stop the pathogenic events at their initial stages and potentially result in resolution of the pathological process. The rationale for using such an approach can be further substantiated by the fact that Th2 pathway for antibody response is activated and that inhibition of B cells and of pathogenic antibodies is strictly associated with beneficial effects of immunosuppressive drugs in experimental MN.

This is a open-label Phase I/II pilot study. Patients will receive Rituximab at a total dose of 1g on Day 1 and Day 15 according to infusion guidelines. Patient experience complete clinical response (as per response criteria outlined below), AND Patient subsequently experiences clinical relapse, defined as return of proteinuria to 4 g/24h, and in whom CD20+ cell count have normalized, will receive a second course of Rituximab. Patients who relapse but who remain B cell depleted will not be retreated.

ELIGIBILITY:
Patients must meet the following inclusion criteria to be eligible for study entry:

* Membranous Nephropathy with diagnostic biopsy performed within the last 3 years. Renal biopsy slides and electron photomicrographs will be reviewed by study investigators, and must confirm a diagnosis of MN.
* Age  18 years.
* Proteinuria as measured via Uprot/UCr ratio > 4.0 on a spot sample of a 24-hour urine collection, despite ACE inhibitor / ARB treatment. The choice of urine protein/creatinine ratios is in accord with recently developed National Kidney Foundation Chronic Kidney Disease (NKF-CKD) guidelines.107 The NKF-CKD guidelines advocate urine protein/creatinine ratios as the preferred method for evaluation of urinary protein excretion in both adults and children.
* Patients need to be treated with an ACEI and/or ARB, for at least 3 months prior to enrollment with adequately controlled blood pressure (BP <140/80 mm Hg in >75% of the readings).
* Women must be post-menopausal, surgically sterile or practicing a medically approved method of contraception.
* Patients with thromboembolic complications and/or clinical signs of NS that are not controlled with conventional medical treatment will enter the immunosuppressive portion of the protocol (Rituxan treatment) without the 3 months of ACE/ARB treatment (high risk patients).
* Able and willing to give written informed consent and comply with the requirements of the study protocol
* Adequate renal function as indicated by estimated GFR ≥ 25 ml/min per 1.73m2 and/or or serum creatinine <4.0 mg/dL in the presence of ACE inhibitor/ARB therapy. The GFR will be estimated using the 4 variable MDRD equation as published in the NKF-CKD guidelines. The same NKF-CKD guidelines also promote the use of estimated GFR (GFRest) values rather than serum creatinine levels or creatinine clearance measurements as the preferred non-invasive method of determining glomerular filtration rates.107 We have opted to use this approach rather than the much more expensive and more invasive techniques that employ clearance measurements of exogenous substances (such as inulin or iothalamate) since the likelihood of detecting significant changes in GFR in this short term study is remote - no matter which method is chosen. The inclusion of and/or serum creatinine <4.0 mg/dL is to cover possibility of incomplete 24-hour collection at time baseline creatinine clearance.)
* Adequate liver function, as indicated by bilirubin, AST, and alkaline phosphatase levels (up to < 2.5 times the upper normal limit).
* Negative serum pregnancy test (for women of child bearing age)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment or a period of 21 months for those undergoing retreatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-08; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
1. Change from baseline in proteinuria at six and twelve months following treatment
Toxicity/Safety
PK/bioavailability

SECONDARY OUTCOMES:
Partial Remission at 6 months
Complete and Partial Remission at 6 months
Time to CR and time to CR or PR
Rates of decline in GFR and UP

CONTACTS AND LOCATIONS:
Overall Officials: Fernando C. Fervenza, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States